CLINICAL TRIAL: NCT03454035
Title: Ulixertinib (BVD-523) in Combination With Palbociclib in Patients With Advanced Solid Tumors With Expansion Cohort in Previously Treated Metastatic Pancreatic Cancer and Metastatic RAS-mutant and NF1-mutant (no BRAFV600 Mutations) Melanoma
Brief Title: Ulixertinib/Palbociclib in Patients With Advanced Pancreatic and Other Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: BioMed Valley Discoveries, Inc (Industry); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC1736
Record Dates: First submitted 2018-02-05; First posted 2018-03-05 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Tumor, Solid; Pancreatic Cancer; Melanoma
MeSH Terms: conditions — Neoplasms; Pancreatic Neoplasms; Melanoma | interventions — ulixertinib; palbociclib

STUDY DESIGN:
Intervention Model Description: This is a standard 3+3 dose escalation design.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open-label, single arm Phase I (Experimental): Ulixertinib added to palbociclib
  Interventions: Drug: Ulixertinib; Drug: Palbociclib

INTERVENTIONS:
Drug: Ulixertinib — Ulixertinib 300mg, orally, twice a day concomitantly with palbociclib
  Other Names: BVD-523
Drug: Palbociclib — Drug: Palbociclib 125mg, orally, once a day concomitantly with ulixertinib
  Other Names: Ibrance

SUMMARY:
This phase I study is designed to establish the safety, maximally tolerated dose (MTD) and recommended phase II dose (RP2D) of the ERK inhibitor ulixertinib (BVD-523) when combined with the CDK4/6 inhibitor palbociclib.

DETAILED DESCRIPTION:
This phase I study is designed to establish the safety, maximally tolerated dose (MTD) and recommended phase II dose (RP2D) of the ERK inhibitor ulixertinib (BVD-523) when combined with the CDK4/6 inhibitor palbociclib.

Up to a maximum of 30 adult patients will be enrolled in the 5 possible dose escalation cohorts. These patients will have histologically confirmed advanced solid tumor disease refractory to standard of care therapy, or for which there is no accepted standard of care.

An expansion cohort enrollment will start After RP2D of ulixertinib combined with palbociclib is defined. Then 15 patients with metastatic pancreatic cancer and 15 patients with RAS-mutant melanoma will be enrolled.

Note:Pancreatic cancer expansion cohort and all solid tumor cohorts are closed to enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and HIPAA authorization for release of personal health information. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
2. Age ≥ 18 years at the time of consent (no upper age limit)
3. Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 2
4. Tumor Eligibility:

   1. Dose escalation cohorts: Histologically confirmed advanced solid tumor refractory to standard of care therapy, or for which there is no accepted standard of care
   2. Expansion cohort (at RP2D): metastatic pancreatic cancer or malign melanoma patients who have received at least one line of therapy in the metastatic setting
   3. Expansion cohort (at RP2D) for histologically confirmed unresectable stage III or stage IV melanoma with the following additional eligibility requirements:

      * Tumors molecular profiling genetic aberrations: NRASG12/G13/Q61, KRASG12/G13, HRASG12/G13, any amplifications of the NRAS, KRAS, or HRAS genes. For NF1 mutations, subjects with loss-of-function NF1mutations and without any BRAFV600 mutations will be enrolled.
      * Documented disease refractory to at least one PD1/PD-L1 inhibitor, defined as disease progression following at least two infusions of the same drug.
      * Subjects with RAS-mutant and NF1-mutant (no concurrent BRAFV600 mutations) melanoma that have not taken prior immune checkpoint inhibitors will be allowed if they are not eligible to receive prior immune checkpoint inhibitors due to requirement for immunosuppression
5. Measurable or non-measurable (but evaluable) disease according to RECIST v1.1 for dose escalating cohorts; measurable disease as per RECIST v1.1 required for expansion cohort
6. Life expectancy ≥ 12 weeks
7. Recovered from all reversible acute toxic effects of last anti-cancer treatment (other than alopecia) to ≤Grade 1 or baseline. Patients with baseline neuropathy that is ≤ grade 2 are eligible for enrollment.
8. Demonstrate adequate organ function as defined in the table below; all screening labs to be obtained within 28 days prior to day -6 of ulixertinib

   Hemoglobin (Hgb) ≥ 9 g/dL Absolute Neutrophil Count (ANC) ≥ 1,500 /mm3 Platelets ≥ 100,000/mm3 Creatinine ≤1.5 x upper limit of normal (ULN) or Calculated creatinine clearance ≥ 60 mL/min using the Cockcroft-Gault formula Bilirubin ≤ 1.5 x ULN Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤ 2.5 x ULN; if tumor involvement of the liver ≤ 5 x ULN

   *Note: Hematology and other lab parameters that are ≤ grade 2 but still meet the criteria for study entry are allowed. Furthermore, changes in laboratory parameters during the study should not be considered adverse events unless they meet the criteria for dose modification(s) of study medication outlined by the protocol and/or worsen from baseline during therapy.
9. Adequate cardiac function; left ventricular ejection fraction (LVEF) >50% as assessed by ultrasound/echocardiography (ECHO); corrected QT interval (QTc) <470ms
10. Females of childbearing potential must have a negative serum pregnancy test within 3 days prior to day -6 of ulixertinib. NOTE: Females are considered of childbearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are naturally postmenopausal for at least 12 consecutive months
11. Females of childbearing potential and males must be willing to abstain from heterosexual activity* or use effective methods of contraception from the time of informed consent until 120 days after treatment discontinuation. Acceptable contraception methods can be comprised of an intrauterine device (IUD), vasectomy of a female subject's male partner, contraceptive rod implanted into the skin, OR use of two of the following: diaphragm with spermicide (cannot be used in conjunction with cervical cap/spermicide), cervical cap with spermicide (nulliparous women only), contraceptive sponge (nulliparous women only), male condom or female condom (cannot be used together), hormonal contraceptive.] *Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
12. Subject is willing and able to comply with study procedures based on the judgment of the investigator or protocol designee.
13. Willing to provide archival tissue (if available) and consent to mandatory pretreatment and on-treatment biopsy as deemed safe by the treating physician (expansion cohort only) for research purposes only.

Exclusion Criteria:

1. Pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated on the study)
2. Treatment with any cancer-directed therapy (chemotherapy, hormonal therapy, biologic, radiation or immunotherapy, etc.) or investigational drug within 28 days or 5 half-lives (whichever is shorter) prior to day -6 of ulixertinib
3. A history or current evidence/risk of retinal vein occlusion (RVO) or central serous retinopathy (CSR).
4. Major surgery within 28 days prior to day -6 of ulixertinib
5. Not willing to avoid grapefruit, grapefruit juices, grapefruit hybrids, oranges, pummelos, and exotic citrus fruits from 7 days prior to day -6 of ulixertinib and during the entire study due to potential CYP3A4 interaction with the study medications.
6. Intake of any herbal preparations or medications (including, but not limited to, Saint John's Wort and ginkgo biloba) and dietary supplements within 7 days prior to day -6 of ulixertinib due to potential CYP3A4 interaction with the study medications
7. Unable or unwilling to discontinue use of any drug known to be a strong inhibitor of CYP3A4, CYP1A2 or CYP2D6 or strong inducer of CYP3A4 (prohibited inducers and inhibitors must be discontinued within 2 weeks prior to day -6 of ulixertinib; see section 10.3 Appendix C)
8. Unable or unwilling to discontinue use of any drug known to be a sensitive CYP3A4 substrate with a narrow therapeutic index as defined in the protocol.
9. Central nervous system metastases are allowed only for patients RAS-mutated and NF1-mutant melanoma cohorts (1) no leptomeningeal disease is present, (2) Intracranial disease is controlled by prior therapies, as evidenced by brain imaging 2 weeks post treatment indicating no new intracranial disease, (3) stable or decreasing dose of steroids is provided patient on ≤ 20mg of prednisone or it's equivalent daily.
10. Any important medical illness or abnormal laboratory finding that would increase the risk of participating in the study (based on the investigator's judgment)
11. Psychiatric illness/social situations that would limit compliance with study requirements
12. Has a known additional malignancy that is active and/or progressive requiring treatment; non-melanoma skin cancers, non-invasive bladder cancer, and carcinoma in situ of the cervix, prior history of prostate cancer provided the patient is not undergoing active systemic treatment other than hormonal therapy and has documented PSA that is undetectable (<0.2ng/mL), prostate carcinoma in remission and did not receive systemic treatment, papillary thyroid cancer did not receive adjuvant radioactive iodine, Stage Rai stage 0 Chronic lymphocytic leukemia does not require systemic treatment, lymphoma, hairy-cell leukemia, or myelodysplasia is in complete remission and or other cancer for which the patient has been disease-free for at least two years.

    Has a known additional malignancy that is active and/or progressive requiring treatment.
13. Impaired GI function or GI disease that may significantly impair absorption (e.g., inflammatory bowel disease (IBD), malabsorption syndrome, small bowel resection, uncontrolled vomiting or diarrhea)
14. Inability to swallow oral medications
15. Patients with autoimmune diseases that require systemic corticosteroid treatment.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2018-01-30 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-11-24 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Five weeks
  MTD of ulixertinib in combination with palbociclib in patients with advanced solid tumors of ulixertinib in combination with palbociclib in patients with advanced solid tumors
Overall Survival | 6 months after treatment
  For Expansion Cohort: To estimate overall survival (OS) after treatment with the recommended phase 2 dose of ulixertinib in combination with palbociclib in an expansion cohort of patients with metastatic pancreatic cancer

SECONDARY OUTCOMES:
Safety (number of patients with adverse events) | 5 weeks
  Number of patients with adverse events
Objective Response Rate | 8 weeks
  To estimate objective response rate (ORR) after treatment with ulixertinib in combination with palbociclib
Progression-free survival | Up to two years after treatment
  To estimate progression-free survival (PFS) after treatment with ulixertinib in combination with palbociclib
Overall Survival | Up to two years after treatment
  For Expansion Cohort: To estimate overall survival (OS) after treatment with the recommended phase 2 dose of ulixertinib in combination with palbociclib in an expansion cohort of patients with metastatic pancreatic cancer
Cancer Antigen 19-9 (CA19-9) response | Through treatment completion, approximately 1 year
  For Expansion Cohort: To estimate CA19-9 response after treatment with ulixertinib in combination with palbociclib

CONTACTS AND LOCATIONS:
Overall Officials: Stergios Moschos, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States